CLINICAL TRIAL: NCT07369024
Title: Sub-dissociative Dose Ketamine in Treatment of Vaso-occlusive Pain Event in Children and Young Adults: A Randomized Control Trial
Brief Title: Sub-dissociative Dose Ketamine in Treatment of Vaso-occlusive Pain Event in Children and Young Adults
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mohsen Saidinejad (Other)
Responsible Party: Sponsor-Investigator, Mohsen Saidinejad, Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Organization: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-33412-01
Record Dates: First submitted 2026-01-23; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease; Vaso-Occlusive Pain Episode in Sickle Cell Disease; Ketamine Infusion; Pain Management; Vaso-Occlusive Crises
Keywords: Sickle Cell Disease; Vaso-Occlusive Pain Episode; Sub-Dissociative Ketamine; Pediatric Pain Management
MeSH Terms: conditions — Anemia, Sickle Cell; Agnosia; Vaso-Occlusive Crises

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sub-dissociative Ketamine (Experimental): Participants receiving 0.25 mg/kg infusion of ketamine
  Interventions: Drug: Sub-dissociative Ketamine Infusion
- Normal Saline (Placebo Comparator): Participants receiving 100 milliliters of normal saline
  Interventions: Drug: Normal Saline Placebo Infusion

INTERVENTIONS:
Drug: Sub-dissociative Ketamine Infusion — 0.25 mg/kg of IV ketamine within a 20-minute infusion of 100 milliliters of normal saline (NS)
  Arms: Sub-dissociative Ketamine
Drug: Normal Saline Placebo Infusion — 20-minute infusion of 100 milliliters of normal saline
  Arms: Normal Saline

SUMMARY:
The purpose of this research is to see if ketamine is effective and safe in treating children and young adults with sickle cell disease experiencing sickle cell related pain. In this study, we will compare the outcomes (such as pain scores) in persons who receive standard of care pain medicine (an opioid such as morphine) plus a low dose (amount) of ketamine to those who receive only standard of care pain medicine.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages 5-20 years
* Diagnosed sickle cell disease. Homozygous (HbSS) or heterozygous (HbSC, HbSBetaThal Plus or Zero) will be included.
* Presenting with VOE pain, requiring IV pain medication.
* First dose of analgesic medication is given before patient approached for participation in the study.
* Primary language is English or Spanish
* Adult individual or parent/legal guardian is able and willing to provide informed consent. For individuals 7 to 17 years of age, assent must also be provided when cognitively possible.

Exclusion Criteria:

* Sickle cell trait only
* Patients whose primary language is other than English or Spanish
* Pain attributed to causes other than VOE
* Not requiring IV for pain treatment
* No analgesic (e.g. opiate) is given before approach for study participation due to any reason, including problem with IV access.
* Oxygen saturation < 90% on room air
* History of prior adverse reaction to ketamine
* History of hypertension - Patients with active/uncontrolled hypertension defined as systolic 140 mmHg over diastolic of 90 mmHg will be excluded from participation in the study. If hypertension is controlled and at the time of enrollment, systolic and diastolic thresholds of 140 mmHg and 90 mmHg respectively are not exceeded, patient may be included in the study
* History of significant or uncontrolled cardiovascular disease, liver disease, kidney disease, and thyroid disease
* Patients with evidence of increased intracranial pressure
* Patients with elevated intraocular pressure
* Patients with acute mania or history of bipolar disorder with manic episodes, history of hallucinations or paranoia secondary to previously diagnosed psychiatric condition
* Pregnant or potentially pregnant patients per patient report. All patients of childbearing potential will undergo pregnancy testing prior to enrollment (as part of clinical care), and if positive, will be excluded.
* Elevated liver enzymes (alkaline phosphatase, ALT, AST, bilirubin) as sign of hepatic disfunction if the laboratory results are available prior to study participation
* Patients who appear intoxicated on any substance.
* Patients who are wards of the state or prisoners as defined by DHS
* Patients who are not deemed to be competent to provide consent or assent.

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Total Opioid Medications Required for Analgesia | Up to 3 days
  Cumulative morphine-mg equivalent per kilogram (MME/kg) of opioid medication needed to achieve a pain score of ≤ 5

SECONDARY OUTCOMES:
Pain Score | 30 minutes and 60 minutes after administration of placebo vs ketamine infusion
  Pain score from 0-10, at 30 and 60 minutes after administration of NS/placebo (control group), versus sub-dissociative ketamine (experimental group)
ED Length of Stay | Up to 3 days
  To compare ED length of stay between control vs experimental group
Rate of Hospitalization | Up to 1 month
  To compare rate of hospitalization and length of hospitalization between control and experimental group
Quality of Life (Pediatric Quality of Life) | 7-10 days after enrollment in the study and 4-6 weeks after enrollment in the study
  To compare overall quality of life between the two groups upon discharge from the ED or the hospital, using the Pediatric Quality of Life (PedsQL) questionnaire. The questionnaire has 43 points and is reverse scored and linearly transformed to a 0-100 scale (0=100, 1=75, 2=50, 3=25, 4=0), so that higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Harbor UCLA Medical Center, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No